CLINICAL TRIAL: NCT05612919
Title: Safety, Feasibility and Efficacy of Red Blood Cells From Umbilical Cord Blood for Transfusion of Extremely Preterm Infants: Clinical Phase
Brief Title: Red Blood Cells From Umbilical Cord for Transfusion of Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Banc de Sang i Teixits (Other); Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BST-TSCU-01
Record Dates: First submitted 2022-04-05; First posted 2022-11-10 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2023-09

CONDITIONS: Infant, Extremely Premature; Erythrocyte Transfusion; Umbilical Cord Issue
Keywords: Anaemia of prematurity; Extremely preterm infants; Umbilical cord blood; Blood bank; Fetal hemoglobin
MeSH Terms: conditions — Anemia; beta-Thalassemia

STUDY DESIGN:
Intervention Model Description: This is a pilot, open, non-randomized, single-center clinical study, whose main objective is to evaluate the safety, feasibility and efficacy of red blood cell from umbilical cord blood (UCB-RBC) transfusion in extremely preterm infants (EPI).
  When infants fit criteria for red blood cells transfusion the blood bank of reference will be contacted and availability of compatible UCB-RBC bags within those 6 hours will be checked. When it is possible (available compatible UCB-RBC bag within 6 hours), UCB-RBC will be transfused, otherwise patient will receive RBC from adult donor. Patients who initially received RBC from adult donor will remain in this group if repeated transfusions are needed. In patients who initially received UCB-RBC transfusion, availability of compatible UCB-RBC bags will have to be reviewed again. Only when it is not possible to transfuse UCB-RBC at this repeated occasion, the patient will receive RBC from adult blood donor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patients exclusively transfused with UCB-RBC (Experimental): Interventional group infants arm will receive UCB-RBC bag when RBC transfusion is indicated as per standard practice, and when UCB-RBC is available within the first 6 hours of the request.
  Interventions: Other: Red blood cell from umbilical cord blood
- Patients exclusively transfused with AB-RBC (Active Comparator): Standard treatment group infants arm will receive AB-RBC when RBC transfusion is indicated as per standard practice, and compatible UCB-RBC bag is not available.
  Interventions: Other: Red blood cell from adult donor
- Non transfused patients (No Intervention): Patients with no indications for RBC transfusion. Their clinical management will be the usual in our neonatal unit.

INTERVENTIONS:
Other: Red blood cell from umbilical cord blood — Patients will receive a volume of 15-20 ml/kg of red blood cell from umbilical cord blood (UCB-RBC). The transfusion will be prescribed and administered with all the routine safety measures carried out by the nurses to ensure compatibility between the administered RBC and the patient. The UCB-RBC bags will contain a minimum volume of 20 mL of RBC, with a haematocrit of about 60% and an acceptable residual leucocyte content of <106/mm3.
  Product validation is currently under development.
  Arms: Patients exclusively transfused with UCB-RBC
Other: Red blood cell from adult donor — Patients will receive a volume of 15-20 ml/kg of red blood cell from adult donor according to standard guidelines.
  The transfusion will be prescribed and administered with all the routine safety measures carried out by the nurses to ensure compatibility between the administered RBC and the patient.
  Blood samples are irradiated according to standard practise.
  Arms: Patients exclusively transfused with AB-RBC

SUMMARY:
This study has been designed to demonstrate that red blood cell from umbilical cord blood (UCB-RBC) is a safe and available product for extremely preterm infants (EPI) transfusion and that transfusion of UCB-RBC is non-less effective than RBC from adult donor for the treatment of anemia of prematurity in this group of patients.

DETAILED DESCRIPTION:
Prematurity is an important maternal and child health problem due to its incidence and associated complications. Anaemia is a frequent problem in extremely preterm infants (EPI) whose treatment often requires red blood cell (RBC) transfusion. This product is currently obtained from adult blood (AB) donor. The incidence of some prematurity complications have been demonstrated to increase with AB-RBC tranfusions mainly because of the higher oxygen tissue release, such as retinopathy of prematurity (ROP), bronchopulmonary dysplasia (BPD), and necrotizing enterocolitis (NEC). In addition, AB-RBC could contain small amounts of heavy metals that could be toxic for EPI.

RBC from umbilical cord blood (UCB-RBC) might be a better alternative as it does not change the hemoglobin profile and consequently might decrease the oxygen toxicity.

Several studies have evaluated the safety of UCB-RBC transfusions in preterm infants without finding a higher risk of complications compared with AB-RBC transfusions.

A pilot study has been designed to evaluate the safety of UCB-RBC for transfusion in EPI and to determine the feasibility and efficacy of UCB-RBC for transfusion in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from parents or legal guardians
* Preterm infants born earlier than 28 weeks of gestational age.
* Admission to the neonatal intensive care unit of the participating hospital (Hospital Clínic of Barcelona)

Exclusion Criteria:

* Previous transfusion
* Isoimmunization
* Hydrops fetalis
* Major congenital malformations
* Congenital infections
* Hemoglobinopathies
* Extreme urgency of blood availability (hypovolemic shock, disseminated intravascular coagulopathy...)
* Be part of another clinical trial that may interfere with the results

Max Age: 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2023-09-13 (Actual); Primary Completion 2025-07-12 (Actual); Study Completion 2025-07-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with abnormal physical examination after red blood cells from umbilical cord blood (UCB-RBC) transfusion | 24 hours after the procedure
  The number of participants with abnormal physical examination after UCB-RBC transfusion will be analyzed to evaluated the safety of UCB-RBC in extremely preterm infants (EPI)
Number of participants with abnormal vital signs after UCB-RBC transfusion | 24 hours after the procedure
  The number of participants with abnormal physical examination after UCB-RBC transfusion will be analyzed to evaluated the safety of UCB-RBC in EPI
Number of participants with altered value of continous monitoring of regional cerebral and somatic oxygen saturation by near-infrared spectroscopy after UCB-RBC transfusion | 24 hours after the procedure
  The number of participants with Altered value of continous monitoring of regional cerebral and somatic oxygen saturation by near-infrared spectroscopy after UCB-RBC transfusion will be analyzed to evaluated the safety of UCB-RBC in EPI
Number of participants with abnormalities in the result of acid-base balance and ionogram after UCB-RBC transfusion | 24 hours after the procedure
  The number of participants with abnormalities in the result of acid-base balance and ionogram after UCB-RBC transfusion will be analyzed to evaluated the safety of UCB-RBC in EPI
Number of participants with morbidities up to 36 weeks of postmenstrual age after UCB-RBC transfusion | 24 hours after the procedure
  The number of participants with Morbidities up to 36 weeks of postmenstrual age after UCB-RBC transfusion will be analyzed to evaluated the safety of UCB-RBC in EPI

SECONDARY OUTCOMES:
Feasibility of UCB-RBC in EPI | within 6 hours of the request
  Feasibility will be considered proven if UCB-RBC is available in >50% of patients
Total volumen of RBC transfused in transfused patients | An average of 3 month (when patients are 36 weeks of postmenstrual age)
  Total volumen of RBC transfused measured in milliliters will be evaluated to assess the efficacy of UCB-RBC in EPI according to the treatment group (only UCB-RBC, only AB-RBC, both)
Number of RBC tranfusions in transfused patients | An average of 3 month (when patients are 36 weeks of postmenstrual age)
  The total number of RBC transfusions will be evaluated to assess the efficacy of UCB-RBC in EPI according to the treatment group (only UCB-RBC, only AB-RBC, both)
The number of days between two consecutive RBC transfusion in transfused patients | An average of 3 month (when patients are 36 weeks of postmenstrual age)
  The number of days between two consecutive RBC transfusion in each transfused patient will be evaluated to assess the efficacy of UCB-RBC in EPI according to the treatment group (only UCB-RBC, only AB-RBC, both)
Total hemoglobin value (g/dl) in transfused patients | Before transfusion, 24 hours, 1 week, 1 month after transfusion
  Total hemoglobin (g/dl) in transfused patients will be evaluated to assess the efficacy of UCB-RBC in EPI according to the type of transfusion (UCB-RBC vs AB-RBC) An increment in total hemoglobin by 4 ± 2 g / dL 24 hours after the transfusion will be considered significative. Samples will be analysed by microhematocrit method ("Rapidpoint 5000 system, Siemens").
Hematocrit value (%) in transfused patients | Before transfusion, 24 hours, 1 week, 1 month after transfusion
  Hematocrit (%) in transfused patients will be evaluated to assess the efficacy of UCB-RBC in EPI according to the type of transfusion (UCB-RBC vs AB-RBC) An increment in hematocrit by 12 ± 5 points 24 hours after the transfusion will be considered significative. Samples will be analysed by microhematocrit method ("Rapidpoint 5000 system, Siemens").
Fetal haemoglobin value (%) in transfused patients | Before transfusion, 24 hours, 1 week, 1 month after transfusion
  Fetal haemoglobin (%) in transfused patients will be evaluated to assess the efficacy of UCB-RBC in EPI according to the type of transfusion (UCB-RBC vs AB-RBC) A variation of fetal haemoglobin percentage between values before and after the transfusion will be considered significative. It will be analysed by capillary electrophoresis ("Capillary neonatal Hb" kit).
Regional cerebral and somatic oxygen saturation (%) value | Before transfusion, 24 hours, 1 week, 1 month after transfusion
  Regional cerebral and somatic oxygen saturation (%) in transfused patients will be evaluated to assess the efficacy of UCB-RBC in EPI according to the type of transfusion (UCB-RBC vs AB-RBC). Measurements will be taken by near-infrared spectroscopy

OTHER OUTCOMES:
Marrow regeneration | 1 month
  Comparison of reticulocyte counts between transfused and non-transfused patients.
Ferritin value in transfused and non-transfused patients | 1 month
  Ferritin value will be assessed to comparison iron metabolism in transfused and non-transfused patients
Transferrin saturation index (%) in transfused and non-transfused patients | 1 month
  Transferrin saturation index (%) will be assessed to comparison iron metabolism in transfused and non-transfused patients

CONTACTS AND LOCATIONS:
Overall Officials: Miguel María Alsina Casanova, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic of Barcelona, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Widness JA. Pathophysiology of Anemia During the Neonatal Period, Including Anemia of Prematurity. Neoreviews. 2008 Nov 1;9(11):e520. doi: 10.1542/neo.9-11-e520. PMID 20463861
- [Background] Jiramongkolchai K, Repka MX, Tian J, Aucott SW, Shepard J, Collins M, Kraus C, Clemens J, Feller M, Burd I, Roizenblatt M, Goldberg MF, Arevalo JF, Gehlbach P, Handa JT. Lower foetal haemoglobin levels at 31- and 34-weeks post menstrual age is associated with the development of retinopathy of prematurity : PacIFiHER Report No. 1 PacIFiHER Study Group (Preterm Infants and Fetal Haemoglobin in ROP). Eye (Lond). 2021 Feb;35(2):659-664. doi: 10.1038/s41433-020-0938-5. Epub 2020 May 14. PMID 32409707
- [Background] Hellstrom W, Martinsson T, Hellstrom A, Morsing E, Ley D. Fetal haemoglobin and bronchopulmonary dysplasia in neonates: an observational study. Arch Dis Child Fetal Neonatal Ed. 2021 Jan;106(1):88-92. doi: 10.1136/archdischild-2020-319181. Epub 2020 Aug 26. PMID 32847833
- [Background] Teofili L, Papacci P, Orlando N, Bianchi M, Molisso A, Purcaro V, Valentini CG, Giannantonio C, Serrao F, Chiusolo P, Nicolotti N, Pellegrino C, Carducci B, Vento G, De Stefano V. Allogeneic cord blood transfusions prevent fetal haemoglobin depletion in preterm neonates. Results of the CB-TrIP study. Br J Haematol. 2020 Oct;191(2):263-268. doi: 10.1111/bjh.16851. Epub 2020 Jun 8. PMID 32510635
- [Background] Mohamed A, Shah PS. Transfusion associated necrotizing enterocolitis: a meta-analysis of observational data. Pediatrics. 2012 Mar;129(3):529-40. doi: 10.1542/peds.2011-2872. Epub 2012 Feb 20. PMID 22351894
- [Background] Bianchi M, Giannantonio C, Spartano S, Fioretti M, Landini A, Molisso A, Tesfagabir GM, Tornesello A, Barbagallo O, Valentini CG, Vento G, Zini G, Romagnoli C, Papacci P, Teofili L. Allogeneic umbilical cord blood red cell concentrates: an innovative blood product for transfusion therapy of preterm infants. Neonatology. 2015;107(2):81-6. doi: 10.1159/000368296. Epub 2014 Nov 15. PMID 25401961
- [Background] Gonzalez EG, Casanova MA, Samarkanova D, Aldecoa-Bilbao V, Teresa-Palacio M, Busquets EF, Figueras-Aloy J, Salvia-Roiges M, Querol S. Feasibility of umbilical cord blood as a source of red blood cell transfusion in preterm infants. Blood Transfus. 2021 Nov;19(6):510-517. doi: 10.2450/2020.0169-20. Epub 2020 Dec 18. PMID 33370228
- [Background] Bianchi M, Orlando N, Barbagallo O, Sparnacci S, Valentini CG, Carducci B, Teofili L. Allogeneic cord blood red blood cells: assessing cord blood unit fractionation and validation. Blood Transfus. 2021 Sep;19(5):435-444. doi: 10.2450/2020.0138-20. Epub 2020 Nov 3. PMID 33196415
- [Background] Kotowski M, Litwinska Z, Klos P, Pius-Sadowska E, Zagrodnik-Ulan E, Ustianowski P, Rudnicki J, Machalinski B. Autologous cord blood transfusion in preterm infants - could its humoral effect be the kez to control prematurity-related complications? A preliminary study. J Physiol Pharmacol. 2017 Dec;68(6):921-927. PMID 29550804
- [Background] Strauss RG, Widness JA. Is there a role for autologous/placental red blood cell transfusions in the anemia of prematurity? Transfus Med Rev. 2010 Apr;24(2):125-9. doi: 10.1016/j.tmrv.2009.11.003. PMID 20303035